CLINICAL TRIAL: NCT00245557
Title: Nuclear Magnetic Resonance Imaging Study of Treatment With Sertraline in Geriatric Depression
Brief Title: Magnetic Resonance Imaging Study of Geriatric Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Pfizer (Industry); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Brent Forester, Director, Mood Disorders Division, Geriatric Psychiatry Research Program, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004P-002540
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Geriatric; MRI; Sertraline
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Controls (No Intervention): Healthy Controls undergo MRI and neuropsychological testing
- Depressed (Experimental): Depressed subjects receive experimental drug
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Oral Sertraline Dosage started at 25 mg a day, with increases up to maximum dosage strength of 200 mg a day.
  Duration of treatment was 12 weeks.
  Other Names: Zoloft
  Arms: Depressed

SUMMARY:
The purpose of this study was to use Magnetic Resonance Images to further our understanding of predictors and markers of treatment response and non-response in geriatric depression. We hypothesized that concentrations of high energy metabolites would be lower in depressed elderly compared to non-depressed.

ELIGIBILITY:
Inclusion Criteria:

* DSM- IV (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition) diagnostic criteria for major depressive disorder
* Hamilton Depression Scale- 17 item version score of 18 or higher
* Must speak English
* Women must be post-menopausal

Exclusion Criteria:

* A current or pervious psychiatric disorder other than MDD
* A current unstable medical condition
* A pacemaker or metal implant
* History of alcohol or drug dependence or abuse within the past year
* Current prescription of excluded medications
* Use of a drug within the last 30 days that was not approved for use by governmental authorities.
* If you or a family member works at McLean Hospital

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Forester, M.D, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] Harper DG, Joe EB, Jensen JE, Ravichandran C, Forester BP. Brain levels of high-energy phosphate metabolites and executive function in geriatric depression. Int J Geriatr Psychiatry. 2016 Nov;31(11):1241-1249. doi: 10.1002/gps.4439. Epub 2016 Feb 18. PMID 26891040

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls (Baseline): Healthy Controls undergo MRI and neuropsychological testing
- Depressed (Baseline): Depressed subjects receive sertraline open label for 12 weeks beginning at a dosage of 25 mg a day up to a maximum dosage of 200 mg a day.
Period: Overall Study
Arm/Group | Healthy Controls (Baseline) | Depressed (Baseline)
Started | 17 | 26
Completed | 11 | 10
Not Completed | 6 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls (Baseline) | Depressed (Baseline) | Total
Number analyzed (Participants) | 17 | 26 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 11 | 12
  >=65 years | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (4.8) | 69.3 (10.7) | 70.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 9 | 13 | 22
Region of Enrollment [Number; unit: participants]
  United States | 17 | 26 | 43.0

OUTCOME MEASURES:

1. Primary Outcome: HAM-D 17 (Hamilton Depression Rating Scale)
Description: This is a depression severity rating scale measuring symptoms of depression including mood, sleep, appetite, energy, motivation, guilt, suicidal ideation, concentration, physical complaints, paranoia, anxiety, effect on daily functioning and awareness of illness.
  Scale is from 0 (no depression symptoms) up to a maximum of 66 (severe depression symptoms).
Time Frame: baseline at study entry week 0
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Healthy Controls (Baseline) | Depressed (Baseline)
Number analyzed (Participants) | 11 | 10
Units on a scale | 1.0 (1.1) | 18.5 (6.5)

2. Primary Outcome: Geriatric Depression Scale
Description: This is a depression severity rating scale measuring symptoms of depression. Scale is from 0 (no depression symptoms) up to a maximum of 15 (severe depression symptoms).
Time Frame: baseline at study entry week 0
Population: Not all subjects included in MRS analysis had baseline GDS data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Healthy Controls (Baseline) | Depressed (Baseline)
Number analyzed (Participants) | 10 | 9
Units on a scale | 0.6 (.51) | 9.1 (1.6)

3. Primary Outcome: Phosphorus Magnetic Resonance Spectroscopy (31P-MRS)
Description: The primary outcome is a phosphorus magnetic resonance spectroscopy (31P-MRS) signal quantified using a spectral time-domain fitting program based on the Marquadt-Levenberg non-linear, least-squares algorithm, that incorporates prior knowledge of spectral peak assignments, chemical shifts and J-coupling constants. Least squares means were calculated for average total signal using linear mixed effects models. Results are expressed as a spectroscopic index.
  beta-nucleoside triphosphate (bNTP) Phosphocreatine (PCr) Total nucleoside triphosphate (NTP)
Time Frame: at week 0 for both control and depressed, and at week 12 for depressed
Measure: Least Squares Mean (Standard Error); unit: Spectroscopic Index
Arm/Group | Healthy Controls (Baseline) | Depressed (Baseline) | Post-treatment Depressed
Number analyzed (Participants) | 10 | 9 | 8
Spectroscopic Index
  bNTP | .0432 (.0007) | .0397 (.0006) | .0410 (.0007)
  PCr | .0496 (.0009) | .0512 (.0008) | .0515 (.0009)
  Total NTP | .1509 (.0028) | .1420 (.0029) | .1396 (.0028)

ADVERSE EVENTS:
Time Frame: 6 years, 2 months
Arm/Group | Healthy Controls (Baseline) | Depressed (Baseline)
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/26
Other Adverse Events (participants affected / at risk) | 0/17 | 4/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Controls (Baseline) (N=17) | Depressed (Baseline) (N=26)
Loose stools/ Diahrrea (Gastrointestinal disorders) | 0 (0) | 4 (11)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry Mouth (General disorders) | 0 (0) | 3 (5)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Blurred Vision (Eye disorders) | 0 (0) | 2 (2)
Headaches (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No